CLINICAL TRIAL: NCT04495634
Title: Evaluation of a Carbon Nanotube Enabled Solid-State Head CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-0614; W81XWH1820043 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2020-07-28; First posted 2020-08-03 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-08

CONDITIONS: Head Trauma
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Head Trauma or Brain Bleed (Experimental): Medically stable patients who have undergone conventional head CT imaging undergo imaging within 24 hours using the s-HCT system.
  Interventions: Device: Stationary Head CT (s-HCT)

INTERVENTIONS:
Device: Stationary Head CT (s-HCT) — The system consists of a total of three x-ray sources and nine x-ray detectors with an estimation of approximately 150 projection angles per slice, with less than a minute per slice reconstruction. Radiation dose will be configured as to not exceed that of a conventional head CT, or 2 mSv. The subjects will be positioned on a medical procedure table that will move the subject through the scanning system at the rate of roughly 1 cm per second, during which the necessary x-ray projections will be acquired. The head will be positioned in a carbon fiber head holder from a clinical CT scanner that is secured to the table.

SUMMARY:
Purpose: The purpose of this study is to evaluate stationary head CT (s-HCT) as a diagnostic tool in patients with known head trauma.

Participants: Participants will be 50 people who have had either a head trauma or a brain bleed and have undergone a head CT in the past 24 hours or who will undergo a CT scan of the head.

Procedures (methods): This investigation will be a single arm, prospective clinical trial. Participants will have one single visit, which will include the s-HCT scan. No follow-up is required. All images will be de-identified before inclusion within a reader study. The investigators will perform a reader study with physician readers comparing the acquired imaging s-HCT images and conventional head CT.

DETAILED DESCRIPTION:
This investigation will be a single arm, prospective clinical trial evaluating stationary head CT (s-HCT) as a diagnostic tool in patients with known head trauma. The investigators hypothesize that a stationary head CT (s-HCT) system based on the carbon nanotube linear array x-ray source can provide diagnostic quality head CT images. Patients included in the study will be 50 people who have had either a head trauma or a brain bleed and have undergone a head CT in the past 24 hours or who will undergo a CT scan of the head.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Medically stable patient with head trauma or known intracranial hemorrhage (subdural or intraparenchymal) or skull fractures
* Patient has undergone conventional head CT imaging at UNC hospitals within the past 24 hours or will undergo a CT scan of the head
* Willing and able to provide written informed consent

Exclusion Criteria:

* Unable to provide consent
* Any woman who is pregnant or has reason to believe she is pregnant (the possibility of pregnancy has to be excluded by negative urine β-HCG results, obtained within 24 hours prior to the research scan, or on the basis of patient history, e.g., tubal ligation, hysterectomy or a minimum of 1 year without menses)
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Zamora, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Head Trauma or Brain Bleed
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Head Trauma or Brain Bleed
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Stationary Head CT for the Detection of a Hemorrhage
Description: Sensitivity of stationary head CT for the detection of a hemorrhage using a reader study is defined as the ability of readers (radiologists) to use the stationary head CT to predict hemorrhage using conventional head CT as the gold standard. All stationary head CT scans will be reviewed in a standardized reader study at the conclusion of all study imaging.
Time Frame: Upon completion of all study image data collection for all participants [each participant was assessed approximately 1 hour for the duration of the single one-hour visit]
Measure: Mean (Standard Deviation); unit: percent accurately predicted
Units Other Than Participants: CT Scans
Arm/Group | Head Trauma or Brain Bleed
Number analyzed (Participants) | 17
Number analyzed (CT Scans) | 17
percent accurately predicted | 33 (29)
Statistical Analysis 1: Comparison: Head Trauma or Brain Bleed; Test type: Equivalence — The equivalence margin was defined through power calculations based on sample size, power of 0.90 and alpha of 0.05 resulting in a margin of +/- 0.26; p < 0.0001, ANOVA

2. Primary Outcome: Specificity of Stationary Head CT for the Detection of a Hemorrhage
Description: Specificity of stationary head CT for the detection of a hemorrhage using a reader study is defined as the ability of readers (radiologists) to use the stationary head CT to distinguish between individuals that do not have a hemorrhage using conventional head CT as the gold standard. All stationary head CT scans will be reviewed in a standardized reader study at the conclusion of all study imaging.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent accurately identified
Units Other Than Participants: CT Scans
Arm/Group | Head Trauma or Brain Bleed
Number analyzed (Participants) | 17
Number analyzed (CT Scans) | 17
percent accurately identified | 98 (4)
Statistical Analysis 1: Comparison: Head Trauma or Brain Bleed; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.41, ANOVA

3. Primary Outcome: Sensitivity of Stationary Head CT for the Detection of a Fracture
Description: Sensitivity of stationary head CT for the detection of a fracture using a reader study is defined as the ability of readers (radiologists) to use the stationary head CT to predict a fracture using conventional head CT as the gold standard. All stationary head CT scans will be reviewed in a standardized reader study at the conclusion of all study imaging.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent accurately predicted
Units Other Than Participants: CT Scans
Arm/Group | Head Trauma or Brain Bleed
Number analyzed (Participants) | 17
Number analyzed (CT Scans) | 17
percent accurately predicted | 32 (16)
Statistical Analysis 1: Comparison: Head Trauma or Brain Bleed; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0001, ANOVA

4. Primary Outcome: Specificity of Stationary Head CT for the Detection of a Fracture
Description: Specificity of stationary head CT for the detection of a fracture using a reader study is defined as the ability of readers (radiologists) to use the stationary head CT to distinguish between individuals that do not have a fracture using conventional head CT as the gold standard. All stationary head CT scans will be reviewed in a standardized reader study at the conclusion of all study imaging.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent accurately identified
Units Other Than Participants: CT Scans
Arm/Group | Head Trauma or Brain Bleed
Number analyzed (Participants) | 17
Number analyzed (CT Scans) | 17
percent accurately identified | 16 (10)
Statistical Analysis 1: Comparison: Head Trauma or Brain Bleed; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0001, ANOVA

ADVERSE EVENTS:
Time Frame: Each participant assessed for AE's from the time of signing informed consent through the end of the single one-hour visit.
Arm/Group | Head Trauma or Brain Bleed
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT04495634/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT04495634/ICF_001.pdf